CLINICAL TRIAL: NCT00488527
Title: Multicentric, Open Label Clinical Trial. Use of Optimal Method to Initiate and Maintain Lantus Therapy (Insulin Glargine) in Combination With Hypoglycemic Agents, Assessing the Resulting Metabolic Control and the Safety in T2 Diabetes Mellitus Patients.
Brief Title: DOMME Dose Optimization Multicentric Mexican Evaluation
Acronym: DOMME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_01890
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin glargine — Patients will begin with a fixed, subcutaneous dose of insulin glargine, (10 U), in its commercial presentation, which will be adjusted week by week, according to the values of the glycemia when fasting (FBG), adding 2, 4, 6 or 8 units of insulin glargine over the following twelve weeks, during which the therapeutic objective should be attained, namely the glucose goal during fasting of 100 mg/dl (<6.0 mmol/L), and the active treatment is to be continued for three more months.

SUMMARY:
To evaluate the efficiency of Lantus plus combined oral hypoglycaemic agents in terms of respondents percentage. The respondent is defined as the person achieving a value in the final determination of HbA1c < 7% as its absolute value and/or a decreasing in the final value of HbA1c of more than 12% compared with the initial value (final HbA1c vs. initial HbA1c).

Describe the glycemia levels and body weight change in the two response groups, (respondents and non-respondents).

Describe the adverse events Evaluate the safety of using the medication according to the incidence and relevance of the hypoglycemia events, (symptomatic, diurnal, nocturnal, severe).

Estimate the intra-patient variability of the fasting glycemia

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus receiving antidiabetic treatment (1 or 2 oral agents) during more than 6 months, who need a prolonged action basal insulin to control hyperglycemia
* Glycosylated hemoglobin > 8,0% and < 10 %
* Body mass index (BMI) < 40 kg/m2
* Voluntary acceptation of the treatment and capability to self inject the insulin glargine
* Capability and desire to carry out self-determination of glycemia levels using glucometers

Exclusion Criteria:

* Renal function disorder, revealed by a serum creatinine > 177 µmol/l (> 2,0 mg/dl) in Visit 1 or currently undergoing kidney dialysis
* Acute metabolic acidosis (> 1 episode during the last year) or chronic, including diabetic ketoacidosis
* Clinical evidence of an active liver disease or serum ALT/AST >2.5 times the upper normality limit
* A history of unnoticed hypoglycemia
* Surgical treatment for diabetic retinopathy, (laser photocoagulation or a vitrectomy), during the three months prior to joining the trial, or patient that has needed treatment within three months of entering the trial
* Pregnancy or breast feeding
* Not using an adequate birth control method, (only for potentially fertile females) : for example, the use of systemic hormones, (pills or birth control implants), intrauterine devices or a barrier method, (diaphragm with intra-vaginal spermicides, male or female preservative)
* Known hypersensitivity to insulin glargine or any of its excipients
* Malignant process, except for basal carcinoma cells during the last five years
* More than two weeks of continuous treatment with systemic glucocorticoids in the last 6 months
* Concomitant treatment with non-cardio selective beta blockers
* Known supra-renal failure
* Known hemoglobinopathy or anemia, uncontrolled or unstable
* A psychiatric disturbance which prevents the patient from understanding the nature, objective and possible consequences of the trial
* A history of drug or alcohol abuse in the last two years or any current addiction
* Current use of insulin glargine
* Any clinically relevant, cardiovascular, hepatic, neurological, endocrinal or systemic major disease, or any other type, which may hinder the development of the protocol or the interpretation of the results of the trial
* Known existence of GAD (glutamic acid decarboxylase) antibodies
* Type 1 diabetes mellitus, according to its definition by the WHO
* The use of a drug being researched other than insulin during six months prior to joining the trial or the use of an insulin under study during four weeks before entering the trial
* A history of severe hypoglycemia with repeated blackouts, (more than 1), during the last year

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in the initial vs. final values of HbA1c | 9 months
Number of severe hypoglycemia | 9 months

SECONDARY OUTCOMES:
- Change in the fasting glucose values with each visit | 9 months
- Incidences of symptomatic and asymptomatic nocturnal hypoglycemia - Evaluations of safety with regards to the use of insulin glargine, recording the adverse events, excluding hypoglycemia - Abnormal laboratory results | 9 months
- Change in body weight initial visit vs. final visit | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Ruiz, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, México, Mexico